CLINICAL TRIAL: NCT04327583
Title: Pharmaceutical Intervention in the Coordinated Care Pathway for Cancer Patients Treated With Oral Therapy
Brief Title: Impact of the Coordinated Intervention of the Healthcare Facilities Pharmacist and the Dispensary Pharmacist on the Care Pathway for Cancer Patients Treated With Oral Therapy
Acronym: IPPACTTO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ICO-2019-07
Record Dates: First submitted 2020-03-13; First posted 2020-03-31 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Advanced or Metastatic Solid Tumor; Relapsed Hematologic Malignancy
Keywords: Anti cancer oral therapy; Pharmaceutical intervention; Adverse events; Drug interactions; Coordinated care pathway; Drug related problem; Adherence; Quality of life; Pharmaceutical care; Clinical pharmacy; Oncology pharmacy; Hospital pharmacist; Patient satisfaction; Patient care team; Community pharmacist
MeSH Terms: conditions — Neoplasm Metastasis; Hematologic Neoplasms; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coordinated pharmaceutical path (Experimental): Patients treated with anti-cancer oral therapy who benefit a specific pharmaceutical follow-up by the healthcare facilities pharmacist and by the dispensary pharmacist
  Interventions: Behavioral: IPPACTTO
- Standard of care (No Intervention): Patients treated with anti-cancer oral therapy who who do not benefit from an additional pharmaceutical intervention

INTERVENTIONS:
Behavioral: IPPACTTO — The coordinated experimental pharmaceutical path consists of 7 pharmaceutical interviews or consultations. One initial pharmaceutical consultation with the hospital pharmacist. Five follow-up pharmaceutical interviews with the dispensary pharmacist. One follow-up pharmaceutical consultation with hospital pharmacist.
  Each pharmaceutical interview or consultation will result in the drafting of a pharmaceutical report to be sent to the other participating health professionals. At each pharmaceutical consultation or interview, the pharmacists requested perform a clinical pharmaceutical analysis of drug prescriptions; Evaluate the patient's understanding; Detect adherence problems, Identify drug related problems; Alert the oncologist and / or the attending physician.
  Arms: Coordinated pharmaceutical path

SUMMARY:
The rise of oral therapies in the management of cancers has considerably changed the patient care path. If the oral route is preferred by patients because it offers a better quality of life, it is not without impact for patients and the health professionals involved in their management in their care. Indeed, the use of the oral route shifts part of the responsibility for monitoring treatment towards the patient, thereby leading to compliance problems, drug interactions and the management of adverse effects.These risks can cause complications or compromise the effectiveness of treatment, and generate additional costs for the investigator's health system. The study proposes to involve Healthcare Facilities Pharmacist and the Dispensary Pharmacist with all other health professionals.First, the hospital pharmacist will operate before the initiation of an oral route to perform a clinical pharmaceutical analysis of drug prescriptions. Then after the primary prescription and finally during a follow-up consultation 3 months after the initiation of treatment. The hypothesis of the study is that the coordinated intervention of the hospital pharmacist and of the dispensary pharmacist would improve the tolerance of oral treatments by reducing the number of serious adverse effects found, as well as improve the, quality of life, patient and professional satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years old or more
* Having given his written consent to participate in the study
* Patients with advanced or metastatic solid tumor or relapsed hematologic malignancy
* With an initiation of oral therapy
* Performance Status 0, 1 or 2

Exclusion Criteria:

* Patient receiving ongoing intravenous (IV) or subcutaneous (SC) anticancer treatment
* Patient receiving ongoing oral therapy
* Patient receiving first-generation hormone therapy
* Patient receiving ongoing a coordinated pharmaceutical path
* Patient participating in a therapeutic education program including a pharmacist
* Patient already included in an interventional clinical trial
* Oral therapy with Temporary Authorisation
* Patient in a health or medico-social institution
* Patient protected, under guardianship or unable to give free and informed consent
* Patient does not speak French
* Patient unable to read French
* Patient unable to undergo the medical monitoring of the trial for geographical, social or psychological reasons.
* Patients 70 years old with cognitive disorders identified by the G-CODE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Impact of the coordinated pharmaceutical path on the tolerance of oral therapies against cancer. | 6 months from the treatment initiation
  The impact on tolerance will be measured by the proportion of patients with at least one grade 3 or 4 adverse event occurring / confirmed, linked to oral therapy, and confirmed by the oncologist.

SECONDARY OUTCOMES:
Impact of the coordinated pharmaceutical path on the number of grade 3 and 4 adverse events detected linked to oral therapy | 6 months from the treatment initiation
  The impact will be measured by the number of grade 3 and 4 adverse events occurring / confirmed, linked to oral therapy, and confirmed by the oncologist.
Impact of the coordinated pharmaceutical path on unplanned hospitalizations related to the oral therapy | 6 months from the treatment initiation
  Number of unplanned hospitalizations related to the oral therapy and confirmed by the oncologist.
Impact of the coordinated pharmaceutical path on the drug related problems. | 6 months from the treatment initiation
  Number and nature of potential and confirmed drug related problemS detected by pharmacists
Detection of concerted treatment modifications between oncologist and pharmacist related to oral therapy | 6 months from the treatment initiation
  Number of treatment modifications related to oral therapy, necessary before starting treatment and during oral therapy and confirmed by the oncologist during follow-up consultations
Impact of the coordinated pharmaceutical path on quality of life: EORTC QLQ-C30 questionnaire | Inclusion ; 1 month ; 3 months and 6 months from the treatment initiation
  Quality of life for patients will be evaluated by a questionnaire before and after starting oral therapy according to the The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire
Impact of the coordinated pharmaceutical path on adherence to the oral therapy | 1 month ; 3 months and 6 months from the treatment initiation
  Adherence to the oral therapy measured with the Girerd questionnaire wich is composed of 6 questions with an expected answer yes or no. A "yes" answer is worth 1, "No" answer is worth 0. The maximum score obtained is 6; the minimum score is 0. Final Score> 2: low compliance ; Final score = 1 or 2: average compliance ; Final score = 0: good compliance.
Satisfaction of patients related to the coordinated pharmaceutical path: questionnaire | 6 months from the treatment initiation
  Satisfaction of patients will be evaluated by a series of questions related to oral therapy. The patient responds if he strongly disagrees; rather disagree; somewhat agree ; Totally agree. An overall score is also required between 1 and 10; 1 is very bad; 10 is perfect
Assessment of the link between hospital and city | Through study completion, an average of 42 months
  Evaluation of the link will be performed by a questionnaire to be completed by the oncologist and pharmacists. Each responds if he strongly disagrees; rather disagree; somewhat agree ; Totally agree

CONTACTS AND LOCATIONS:
Overall Officials: Fanny D'ACREMONT-JUTIER, Principal Investigator — OMEDIT Pays de la Loire
Locations (7):
- France (7):
  - Institut de Cancérologie de l'Ouest, Angers
  - CHU, Angers
  - Ch Cholet, Cholet
  - CHD Vendée, La Roche-sur-Yon
  - Ch Le Mans, Le Mans
  - Chu Nantes, Nantes
  - Institut de Cancérologie de l'Ouest, Saint-Herblain